CLINICAL TRIAL: NCT00818857
Title: Primary Care Based Randomized Trial to Reduce Cancer Screening Disparities
Acronym: Get Screened
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Kevin Fiscella, Principal Investigator, University of Rochester
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: RSRB 00025557
Record Dates: First submitted 2009-01-06; First posted 2009-01-08 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Preventive Measures
Keywords: cancer screening; screening disparities; underserved populations
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Early intervention.
  Interventions: Behavioral: Early Intervention
- 2 (Active Comparator): Delayed intervention
  Interventions: Behavioral: Delayed intervention

INTERVENTIONS:
Behavioral: Early Intervention — At the point of randomization the early group will receive increasingly intensive reminders to complete specific cancer screening tests.
  Arms: 1
Behavioral: Delayed intervention — One year from the point of randomization patients will begin to receive increasingly intensive reminders to complete specific cancer screening tests.
  Arms: 2

SUMMARY:
The purpose of this project is to improve cancer screening rates within practices serving low-income minority patients

DETAILED DESCRIPTION:
This project is designed to implement and rigorously evaluate a cancer screening quality improvement project within a practice serving underserved patients. The project involves use of a patient registry coupled with patient reminders,recall and outreach.All unscreened patients will receive the benefit of this intervention, though some sooner than others for the purpose of evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Men age 50-75 yrs.
* Women age 40-75 yrs
* One primary care visit in past 2 years.

Exclusion Criteria:

* High risk for colorectal or breast cancer.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1072 (Actual)
Dates: Start 2009-01; Primary Completion 2012-10 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
To test for differences in rates of screening between the early intervention and delayed groups, the chi-square test will be used for each outcome. | End of project, 12/2011

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Fiscella, MD, MPH, Principal Investigator — University of Rochester

REFERENCES:
- [Derived] Fiscella K, Humiston S, Hendren S, Winters P, Idris A, Li SX, Ford P, Specht R, Marcus S. A multimodal intervention to promote mammography and colorectal cancer screening in a safety-net practice. J Natl Med Assoc. 2011 Aug;103(8):762-8. doi: 10.1016/s0027-9684(15)30417-x. PMID 22046855
- [Derived] Fiscella K, Yosha A, Hendren SK, Humiston S, Winters P, Ford P, Loader S, Specht R, Pope S, Adris A, Marcus S. Get screened: a pragmatic randomized controlled trial to increase mammography and colorectal cancer screening in a large, safety net practice. BMC Health Serv Res. 2010 Sep 23;10:280. doi: 10.1186/1472-6963-10-280. PMID 20863395